CLINICAL TRIAL: NCT06448026
Title: Cemiplimab and Cetuximab Prior Salvage Surgery in Patients With Recurrent Oral Cavity Squamous Cell Carcinoma (OCSCC).
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0053; NCI-2024-04824 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Locally Recurrent Oral Cavity Squamous Cell Carcinoma
Keywords: local recurrence; oral cavity cancer
MeSH Terms: conditions — Mouth Neoplasms | interventions — cemiplimab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cemiplimab + Cetuximab (Experimental): Participants will receive cemiplimab and cetuximab together for 6 weeks, and then you will have salvage surgery. Based on how the tumor responds to the study therapy, you may also receive cemiplimab alone for up to 1 year after surgery.
  Interventions: Drug: Cemiplimab; Drug: Cetuximab

INTERVENTIONS:
Drug: Cemiplimab — Given by IV
Drug: Cetuximab — Given by IV

SUMMARY:
To learn if giving cemiplimab and cetuximab before salvage surgery can help to control recurrent oral cavity squamous cell carcinoma.

DETAILED DESCRIPTION:
Primary Objective:

- To assess the efficacy of cemiplimab and cetuximab in patients with recurrent oral cavity squamous cell carcinoma

Secondary Objective:

* To assess safety of cemiplimab and cetuximab prior salvage surgery
* To evaluate the efficacy of cemiplimab and cetuximab prior salvage surgery on measures
* To estimate the one-year disease free survival (DFS)
* To estimate the median overall survival (OS)

Tertiary/Exploratory Objective:

* To explore patient-reported outcomes (PRO) during CC and following salvage surgical resection
* Assess impact of cemiplimab and cetuximab on surgery and adjuvant therapy
* To explore biomarkers that may predict response to therapy

ELIGIBILITY:
Inclusion Criteria:

1. Participants ≥18 years with histology-proven recurrent oral cavity squamous cell carcinoma.
2. Amenable to salvage surgery
3. Disease recurrence at least 3 months after completion of curative-intent therapy (including surgery, post operatory radiation, and/or chemotherapy)
4. Measurable disease per RECIST 1.1
5. Performance status ECOG of 0 or 1
6. Willing to undergo baseline (if archival tumor specimen is not available) and on-treatment biopsy for correlative studies
7. Laboratory measurements, blood counts:

   1. Hemoglobin ≥ 9 g/dL. Red blood cell transfusions are permitted to meet the hemoglobin inclusion criteria
   2. Absolute neutrophil count ≥ 1 x 109/mL
   3. Platelets ≥ 80 x 109/mL
8. Laboratory measurements, renal function:

   a) Creatinine clearance ≥ 30 mL/min as assessed by the Cockcroft-Gault equation
9. Laboratory measurements, hepatic function:

   1. AST and ALT ≤ 3 x ULN
   2. Total bilirubin ≤ 1.5 x ULN or ≤ 3.0 x ULN and primarily unconjugated if subject has a documented history of Gilbert's syndrome or genetic equivalent
10. Female participants with reproductive potential must practice two effective contraceptive measures for the duration of study drug therapy and for at least 90 days after completion of study therapy. The two birth control methods can be either two barrier methods or a barrier method plus a hormonal method to prevent pregnancy. The following are considered adequate barrier methods of contraception: diaphragm, condom, copper intrauterine device, sponge, or spermicide. Appropriate hormonal contraceptives will include any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent (including oral, subcutaneous, intrauterine, or intramuscular agents).
11. Male participants who are sexually active with women with reproductive potential must agree to use contraception for the duration of treatment and for at least 90 days after completion of study therapy.

Exclusion Criteria:

1. Disease recurrence within 3 months after completion of definitive treatment (including surgery, post operatory, systemic therapy)
2. Distant metastatic disease (M1), visceral and/or distant nodal
3. Any prior treatment with an anti-PD1/PD-L1 agent
4. Participants with a condition requiring corticosteroid therapy (>10 mg prednisone/day or equivalent) within 14 days of the first dose of study drug.

   Exceptions: Physiologic replacement doses are allowed even if they are >10 mg of prednisone/day or equivalent, as long as they are not being administered for immunosuppressive intent. Inhaled or topical steroids are permitted, provided that they are not for treatment of an autoimmune disorder.
5. Participants with active, known, or suspected autoimmune disease that has required systemic therapy within 5 years of the projected enrollment date.

   Exceptions: Participants with vitiligo, type I diabetes mellitus, and endocrinopathies (including hypothyroidism due to autoimmune thyroiditis) only requiring hormone replacement, childhood asthma that has resolved, or psoriasis that does not require systemic treatment are permitted.
6. History of interstitial lung disease (eg, idiopathic pulmonary fibrosis, organizing pneumonia) or active, noninfectious pneumonitis that required immune-suppressive doses of glucocorticoids to assist with management.
7. Recipient of a solid organ transplant (other than corneal transplants)
8. Prior allogeneic stem cell transplantation, or autologous stem cell transplantation
9. History of previous malignancy other than malignancy treated with curative intent within less than 5 years. Participants with the following diagnoses represents an exception and may enroll if ≥ 1 year with no evidence of active disease before the first dose of the study drug:

   1. Locally advanced non-melanoma skin cancers with no current evidence of disease
   2. Melanoma in situ with no current evidence of disease
   3. Localized cancer of the prostate with prostate-specific antigen of <1 ng/mL
   4. Treated or localized well-differentiated thyroid cancer
   5. Treated cervical carcinoma in situ
   6. Treated ductal/lobular carcinoma in situ of the breast
10. Evidence of uncontrolled, active infection, requiring systemic anti-bacterial, anti-viral or anti-fungal therapy ≤ 10 days prior to administration of cemiplimab and cetuximab. Subjects with known hepatitis B, hepatitis C (HCV), or HIV infection could go on study if the viral load is undetectable at screening.
11. Disease or medical conditions that would substantially increase the risk-benefit ratio of participating in the study that include acute myocardial infarction within the last 6 months, unstable angina, uncontrolled diabetes mellitus, significant active infections, and congestive heart failure New York Heart Association Class III-IV
12. Female participants who are pregnant or breast-feeding
13. Known hypersensitivity to any of the study drugs, the metabolites, or formulation excipient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2024-11-21 (Actual); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-05-15 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Renata Ferrararotto, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org